CLINICAL TRIAL: NCT06160830
Title: Effects of Synbiotic Supplement on Anthropometric Parameters, Cardiovascular Disease Risk Factors, and Bone Metabolism Markers in Transplanted Kidney Patients on Chronic Post-kidney Transplant Phase Diet
Brief Title: The Effects of Synbiotic on Cardiovascular and Bone Metabolism Markers in Transplanted Kidney Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, zahra yari, faculty, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 051
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Transplanted Kidney
MeSH Terms: interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- synbiotic (Active Comparator): Patients in the synbiotic group will receive, for 10-12 weeks, Two capsules of synbiotic (Zist Takhmir Company) per day, each containing 500 mg of synbiotic. Patients in this group received a multispecies probiotic product (109 CFU/capsule) and fructo oligosaccharid as prebiotics.
  Interventions: Dietary Supplement: synbiotic
- placebo (Placebo Comparator): Patients in the placebo group will receive Two capsules of placebo containing maltodextrin per day. The placebo powder will comparable in color, texture, and taste to the synbiotics. Supplement packaging will be done by Zist Takhmir Company.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: synbiotic — Two capsules of synbiotic per day, each containing 500 mg of synbiotic
  Arms: synbiotic
Other: placebo — Two capsules of placebo containing maltodextrin per day
  Arms: placebo

SUMMARY:
The aim of this double-blind randomized clinical trial is to determine the effects of synbiotic supplement on cardiovascular disease risk factors and bone metabolism markers and depression, in transplanted kidney patients on chronic post-kidney transplant phase diet.This study is a double-blind, randomized controlled clinical trial with two parallel groups. 44 patients will be randomly assigned into synbiotic and control group. Transplanted kidney patients referring to the hospital clinics will be invited to participate. After assessing the entrance criteria, 7 cc blood samples are taken. The food recall is completed. Supplements are given to patients for 10-12 weeks. Serum concentrations of malondialdehyde; high sensitivity c-reactive protein; Soluble intercellular adhesion molecule-1; glucose; pentosidine; carboxy-methyl lysine; osteoprotegerin; Receptor activator of nuclear factor kappa-Β ligand; N-telopeptide; Intact parathyroid hormone; triglyceride; total cholesterol; High-density lipoprotein cholesterol; low-density lipoprotein cholesterol; lipoprotein-a; albumin; calcium; phosphorous; blood nitrogen urea; creatinine; and also systolic blood pressure; diastolic blood pressure; Weight; Body mass index; Waist circumference; Hip circumference; and questionnaires including quality of depression.

ELIGIBILITY:
Inclusion Criteria:

* : More than one year has passed since the last kidney transplant
* Having serum creatinine less than 2.5 mg/dL in the last three months
* Being in the age range of 18-75 years
* BMI<35 kg/m2

Exclusion Criteria:

* Receiving synbiotic supplement

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Lp (a) | 10 weeks
  Serum concentrations of lipoprotein-a
MDA | 10 weeks
  Serum concentrations of malondialdehyde
hs-CRP | 10 weeks
  Serum concentrations of high sensitivity c-reactive protein
sICAM-1 | 10 weeks
  Serum concentrations of Soluble intercellular adhesion molecule-1
glucose | 10 weeks
  serum concentration of fasting glucose
pentosidine | 10 weeks
  serum concentration of pentosidine
carboxy-methyl lysine | 10 weeks
  serum concentration of carboxy-methyl lysine
Osteoprotegerin | 10 weeks
  Serum concentrations of Osteoprotegerin
osteocalcin | 10 weeks
  Serum concentrations of osteocalcin
RANKL | 10 weeks
  Serum concentrations of Receptor activator of nuclear factor kappa-Β ligand
Systolic blood pressure | 10 weeks
  Systolic blood pressure (mmHg)
Diastolic blood pressure | 10 weeks
  Diastolic blood pressure (mmHg)
N-telopeptide | 10 weeks
  Serum concentrations of N-telopeptide
triglyceride | 10 weeks
  Serum concentrations of triglyceride
Total cholesterol | 10 weeks
  Serum concentrations of total cholesterol
HDL-C | 10 weeks
  Serum concentrations of High-density lipoprotein cholesterol
LDL-C | 10 weeks
  Serum concentrations of low-density lipoprotein cholesterol
the Beck depression test | 10 weeks
  Score of the Beck depression test
The Depression Anxiety Stress Scale | 10 weeks
  Score of Depression Anxiety Stress Scale-(DASS)42
Weight | 10 weeks
  body Weight in kilograms
Waist circumference | 10 weeks
  Waist circumference
Hip circumference | 10 weeks
  Hip circumference

SECONDARY OUTCOMES:
albumin | 10 weeks
  Serum concentrations of albumin
calcium | 10 weeks
  Serum concentrations of calcium
phosphorous | 10 weeks
  Serum concentrations of phosphorous
iPTH | 10 weeks
  Serum concentrations of Intact parathyroid hormone